CLINICAL TRIAL: NCT05484050
Title: Estimation of Vascular Endothelial Growth Factor (VEGF) in Iris Tissue in Primary Congenital Glaucoma
Brief Title: VEGF in Iris Tissue in Primary Congenital Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hassan Lotfy Fahmy (Other)
Responsible Party: Sponsor-Investigator, Hassan Lotfy Fahmy, Professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2323300
Record Dates: First submitted 2022-07-22; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Iris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VEGF in iris tissue in primary congenital glaucoma (Other): Estimation of VEGF grade in iris tissue in primary congenital glaucoma through Immunohistochemistry
  Interventions: Other: Immunohistochemistry analysis
- VEGF in iris tissue from ocular trauma or congenital cataract (Other): Estimation of VEGF grade in iris tissue from ocular trauma or congenital cataract through Immunohistochemistry
  Interventions: Other: Immunohistochemistry analysis

INTERVENTIONS:
Other: Immunohistochemistry analysis — Estimation of VEGF through Immunohistochemistry

SUMMARY:
Estimation of vascular endothelial growth factor (VEGF) in iris tissue specimen in primary congenital glaucoma through Immunohistochemistry.

DETAILED DESCRIPTION:
Combined trabeculotomy with mitomycin C will done in infants with primary congenital glaucoma with histopathological examination of the the peripheral iris tissue specimen and vascular endothelial growth factor (VEGF) estimation in iris tissue specimen through Immunohistochemistry.

Estimation of vascular endothelial growth factor (VEGF) in iris tissue specimen taking from ocular trauma or congenital cataract used as control.

ELIGIBILITY:
Inclusion Criteria:

* primary congenital glaucoma

Exclusion Criteria:

* Infants with history of previous surgery.
* Secondary glaucoma.
* Glaucoma associated with other congenital anomalies.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
VEGF | 6 month
  Estimation of VEGF grade in iris tissue through Immunohistochemistry, The grades is arranged from 0 to 5, with 0 being the lowest level and 5 being the highest level

CONTACTS AND LOCATIONS:
Locations (1):
- Hassan Lotfy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No